CLINICAL TRIAL: NCT02191644
Title: Dietary Intervention Replacing Carbohydrate With Protein and Fat Has Greater Effect on Peripheral Blood Mononuclear Cell Metabolites Than on Plasma Metabolites in Patients With Prediabetes or Type-2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PBMC_Lp-PLA2_metabolite
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Prediabetes; Type-2 Diabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Refined rice (Placebo Comparator)
  Interventions: Dietary Supplement: Dietary intervention-refined rice
- Whole grains and legumes (Experimental)
  Interventions: Dietary Supplement: Dietary intervention-whole grains and legumes

INTERVENTIONS:
Dietary Supplement: Dietary intervention-refined rice — Subjects in the control group maintained the usual refined-rice diet.
  Arms: Refined rice
Dietary Supplement: Dietary intervention-whole grains and legumes — Subjects in the whole-grain group replaced refined rice with a mix of 1/3 legumes, 1/3 barley, and 1/3 wild rice three times per day, and increased vegetable intake to at least 6 units (30-70 g/unit) per day for sufficient dietary fiber intake.
  Arms: Whole grains and legumes

SUMMARY:
This study examined whether dietary-induced reductions in lipoprotein-associated phospholipase A2 (Lp-PLA2) activity in peripheral blood mononuclear cells (PBMC) and plasma affected metabolic profiles in PBMCs and plasma.

DETAILED DESCRIPTION:
Eighty nonobese patients (aged 40-70 years) with prediabetes or newly diagnosed type-2 diabetes were randomly assigned to a control group (normal diet with refined rice) or a whole-grain group (replacement of refined rice with whole-grains and legumes). This dietary intervention replaced approximately 7% of carbohydrate-derived energy with approximately 4% of protein-derived energy and approximately 3% of fat-derived energy.

ELIGIBILITY:
Inclusion Criteria:

* subjects who had IFG (100≤ fasting glucose <126 mg/dL)
* or newly diagnosed type-2 diabetes (fasting glucose ≥126 mg/dL)

Exclusion Criteria:

* current and/or past history of cardiovascular disease including angina
* liver or kidney dysfunction
* thyroid or pituitary disease
* pregnancy or lactation
* taking medications or supplements

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Lp-PLA2 Activity in Plasma | Change from baseline in Lp-PLA2 at 12 weeks
Lp-PLA2 Activity in PBMC | Change from baseline in Lp-PLA2 at 12 weeks

SECONDARY OUTCOMES:
PBMC metabolites | Change in L-leucine, oleamide, lysoPC (16:0), and lysoPC (18:0)

OTHER OUTCOMES:
LDL particle size | Changes from baseline in LDL particle size at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Kim M, Song G, Kang M, Yoo HJ, Jeong TS, Lee SH, Lee JH. Replacing carbohydrate with protein and fat in prediabetes or type-2 diabetes: greater effect on metabolites in PBMC than plasma. Nutr Metab (Lond). 2016 Jan 19;13:3. doi: 10.1186/s12986-016-0063-4. eCollection 2016. PMID 26788114